CLINICAL TRIAL: NCT07369479
Title: Effects of a Health Literacy-tailored Self-management Intervention on Blood Pressure Levels Among People With Hypertension: A Randomised Controlled Trial
Brief Title: Effects of a Health Literacy-tailored Self-management Intervention on People With Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hue University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Vo Thi Nhi, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025.809
Record Dates: First submitted 2026-01-13; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hypertension (HTN)
Keywords: hypertension; self-management; health literacy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: health literacy-tailored self-management intervention
- Control group (No Intervention): The participants in the control group will receive care as usual.

INTERVENTIONS:
Behavioral: health literacy-tailored self-management intervention — The participants in the intervention group will receive usual care combine with three weekly face-to-face group sessions (1 hour/week, 6-8 participants) at community health centres, followed by three weekly individual phone call sessions (20 minutes/session).
  Arms: Intervention group

SUMMARY:
This project aims to investigate the effects of a health literacy-tailored self-management intervention among people with hypertension and low health literacy. The primary research question examines the impact of this intervention on blood pressure levels in this population.

Participants will take part in a 6-week intervention consisting of three onsite sessions and three telephone-based sessions, with one session delivered per week. Health literacy-tailored educational materials will be developed to support participants throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Diagnosed with primary hypertension, blood pressure ≥ 140/90 mmHg and taking at least one anti-hypertensive drug
* Health literacy score of 33 or below
* Access to a smartphone
* Able to read and speak in Vietnamese language.

Exclusion Criteria:

* Pregnant women
* Patients with secondary hypertension, psychiatric disorders or cognitive impairments.
* Unable to answer telephone calls.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure levels | Baseline, T1 (immediately post-intervention) and T2 (3 months post-intervention)
  Participants' blood pressure levels will be measured using a validated digital sphygmomanometer.

SECONDARY OUTCOMES:
Proportion of participants achieving optimal blood pressure control | Baseline, T1 (immediately post-intervention) and T2 (3 months post-intervention)
  the number of participants with optimal blood pressure control at each measurement time point divided by the total number of patients enrolled in the group
Medication adherence | Baseline, T1 (immediately post-intervention) and T2 (3 months post-intervention)
  The Vietnamese General Medication Adherence Scale (GMAS) will be used to measure medication adherence across 11 items covering forgetfulness, intentional skipping, complex regimens, and cost-related non-adherence. Items are rated on a 4-point Likert scale from 0 (Strongly disagree) to 3 (Strongly agree), with total scores 0-33; higher scores indicate better adherence. In addition, pill count (the number of pills not used compared to the number of pills received at the most recent prescription filling) will be used as an objective measurement to confirm medication adherence among participants.
Self-management behaviours | Baseline, T1 (immediately post-intervention) and T2 (3 months post-intervention)
  The Vietnamese version of the Hypertension Self-Care Profile Behaviour Scale (HT-SCPB) will be used to measure self-management behaviour. It includes 20 items that address different aspects of self-management behaviour: checking BP, regular visits to doctors, medication adherence, and lifestyle modifications. Each item will be rated on a 4-point Likert scale from 1 (never/rarely) to 4 (always). The total score 20-80, with a higher score indicating higher hypertension self-management behaviours.
Self-efficacy | Baseline, T1 (immediately post-intervention) and T2 (3 months post-intervention)
  The Vietnamese version of the Self-Efficacy for Managing Chronic Diseases (SEM-CD) scale will assess self-efficacy across six items, including confidence in managing fatigue, pain, emotional distress, other symptoms, health-related tasks, and actions beyond medication. Items are rated on a 10-point Likert scale from 1 (not at all confident) to 10 (totally confident), with the mean score (1-10) representing overall self-efficacy.
Health literacy | Baseline, T1 (immediately post-intervention) and T2 (3 months post-intervention)
  The 12-item Vietnamese Short-Form of Health Literacy Questionnaire (HLS-SF12) will be used to measure HL levels (Duong et al., 2019). It includes twelve items that assess how easy it is for patients to find (4 items), understand (3 items), appraise (3 items) and apply health information (2 items). Each item will be rated on a 4-Likert scale (from 1= "Very difficult" to 4="Very easy"). The total score of the scale will be calculated by the formula HL Index = (Mean-1) x (50/3), where Mean is the average score of the 12 items. The HL Index ranges from 0 to 50; a higher score indicates better HL.

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be made available upon reasonable request, subject to ethical approval and data use agreements, to protect participant confidentiality.